CLINICAL TRIAL: NCT06211634
Title: A Phase 1/2, First-in-Human, Single and Multiple Ascending Dose Study to Investigate the Safety, Tolerability, Pharmacokinetics, Pharmacodynamics, and Efficacy of HMB-001 in Participants With Glanzmann Thrombasthenia
Brief Title: A Phase 1/2 Study to Investigate Safety, Tolerability, Pharmacokinetics, Pharmacodynamics, and Efficacy of HMB-001 in Glanzmann Thrombasthenia
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Hemab ApS (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: HMB-001-CL101
Record Dates: First submitted 2024-01-09; First posted 2024-01-18 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-03

CONDITIONS: Glanzmann Thrombasthenia
MeSH Terms: conditions — Thrombasthenia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Single or Multiple ascending dose of HMB-001 (Experimental): Open-label, single or multiple ascending dose of HMB-001
  Interventions: Drug: HMB-001

INTERVENTIONS:
Drug: HMB-001 — HMB-001 is a bispecific antibody being developed as a prophylactic treatment option to prevent and reduce bleeding events in patients with Glanzmann thrombasthenia.

SUMMARY:
The goal of this clinical trial is to Investigate the Safety, Tolerability, Pharmacokinetics, Pharmacodynamics, and Efficacy of HMB-001 in Participants with Glanzmann Thrombasthenia.

The main questions it aims to answer are:

* Parts A, B, and C: To determine the safety and tolerability of HMB-001
* Part A: To establish the dose level(s) and dosing interval(s) of HMB-001 to be investigated in Parts B and C
* Parts B and C: To estimate the ability of HMB-001 to prevent the number and severity of bleeds

Part A will assess differing singular doses of HMB-001 in small groups of participants. The dose administered to a newly enrolled participant (or groups of participants) may only increase if analysis of data from previous dosing shows it is safe to do so. The planned duration of participation in Part A is approximately 6 months, which consists of a Screening Period, an optional Run-in Observation Period, and a follow-up period of 8 weeks.

Part B is similar to Part A as it involves testing different dose levels of HMB-001 in small groups of participants. However, in Part B, HMB-001 is given multiple times over a 3-month period, either weekly, every 2 weeks, or every 4 weeks. Part B consists of a Screening Period, a Run-in Observation Period, a 3-month Treatment Period, and a Safety Follow-up following the last dose of HMB-001.

Part C is open to participants from Part B and consists of approximately a 18-month Treatment Period and a Safety Follow-up following the last dose of HMB-001.

ELIGIBILITY:
Part A Inclusion Criteria:

1. Age 18 to 65 years, at the time of signing informed consent.
2. Glanzmann thrombasthenia; documented abnormal, diagnostic platelet aggregometry plus deficiency of the αIIbβ3 (GPIIb/GPIIIa) receptor via flow cytometry; or genetic diagnosis.
3. Has the ability to provide informed consent.
4. Has an understanding, ability, and willingness to fully comply with trial procedures and restrictions.
5. Vital signs are within the following ranges at Screening:

   1. Resting heart rate ≤ 105 bpm (after at least 5 minutes of resting).
   2. Blood pressure (BP): Resting BP (after at least 5 minutes of resting or based on 24 hours monitor demonstrating normotensive BP): i. Systolic BP: 90 - 140 mmHg. ii. Diastolic BP: 40 - 90 mmHg.
6. Women of child-bearing potential (WOCBP) have a negative serum pregnancy test within 72 hours prior to the first dose of study drug.
7. WOCBP agree to use highly effective contraceptive methods (excluding estrogen-containing combined oral contraceptive pill) as per exclusion criteria and avoid egg donation for 14 days prior to Day 1, during the study treatment, and for 6 months after the last dose of study drug.
8. Men of child-producing potential agree to use highly effective contraceptive methods and avoid sperm donation for 14 days prior to Day 1, during the study treatment, and for 6 months after the last dose of study drug.
9. Participants must meet the following baseline organ function, indicated by laboratory criteria:

   1. Evidence of no greater than mild to moderate reduction in renal function (stage 3a kidney disease), measured by an estimated glomerular filtration rate (eGFR) of ≥45 ml/min/1.73m2 at Screening
   2. An aspartate aminotransferase (AST), alanine aminotransferase (ALT), and total bilirubin ≤ 1.5 x upper limit of normal (ULN) range at Screening. For participants with a history of Gilbert's Syndrome, total bilirubin ≤ 2 × ULN at Screening
   3. Hemoglobin >85 g/L and platelet count >120 x 10^9/L at Screening.

Part B Inclusion Criteria:

1. Has the ability to provide informed consent, and has an understanding, ability, and willingness to fully comply with clinical trial procedures and restrictions.
2. Age 18 to 65 years.
3. Glanzmann thrombasthenia; Genetic diagnosis is required. Abnormal, diagnostic platelet aggregometry plus deficiency of the αIIbβ3 (GPIIb/GPIIIa) receptor via flow cytometry should be recorded if available.
4. Patients should experience bleeding symptoms associated with Glanzmann Thrombasthenia defined as approximately two bleeding events per week of any severity and any type and at least one spontaneous or traumatic bleed that requires a prescribed treatment, medical or surgical procedure within the last 12 months.
5. Vital signs are within the following ranges at Screening:

   1. Resting heart rate ≤105 bpm (after at least 5 minutes of resting)
   2. BP: Resting BP (after at least 5 minutes of resting or based on 24 hours monitor demonstrating normotensive BP): i. Systolic BP: 90 - 140 mmHg; ii. Diastolic BP: 40 - 90 mmHg.
6. Women of child-bearing potential (WOCBP) have a negative serum pregnancy test within 72 hours prior to the first dose of study drug.
7. WOCBP agree to use a highly effective contraceptive method and to avoid egg donation for 14 days prior to Day 1, during the study treatment, and for 6 months after the last dose of study drug. If utilizing an oral contraceptive, women must be on a stable dose of a non-estrogen-containing formulation for at least 8 weeks prior to the start of the Run-in Observation Period and for 8 weeks after the last dose of study drug.
8. Men of child-producing potential agree to use highly effective contraceptive methods and avoid sperm donation for 14 days prior to Day 1, during the study treatment, and for 6 months after the last dose of study drug.
9. Participants must meet the following baseline organ function, indicated by laboratory criteria:

   1. Evidence of no greater than mild to moderate reduction in renal function (stage 3a kidney disease), measured by an eGFR of ≥45 ml/min/1.73m2 at Screening.
   2. An AST, ALT, and total bilirubin ≤1.5 ULN range at Screening. For participants with a history of Gilbert's Syndrome, total bilirubin ≤2 × ULN at Screening.
   3. Hemoglobin >85 g/L and platelet count >120 x 10^9/L at Screening.

Part A Exclusion Criteria

1. Severe infection or inflammation at the time of Screening.
2. History of clinically significant hypersensitivity associated with monoclonal antibody therapies.
3. Personal history of venous or arterial thrombosis or thromboembolic disease, with the exception of catheter-associated, superficial vein thrombosis.
4. Known severe congenital or acquired thrombophilia.
5. Has a positive test for Hepatitis B surface antigen (HbsAg), Hepatitis C antibody (HCV Ab), or human immunodeficiency virus antibody (HIV Ab) at Screening with RNA level above the lower limit of detection. Participants with a positive test for HCV Ab may be included if they have a negative RNA test, consistent with cleared infection. Participants with an HIV RNA level lower than the limit of detection may be included.
6. Other conditions that substantially increase risk of thrombosis by the discretion of the investigator including, but not limited to: significant family history, body mass index (BMI) >30 kg/m2 (moderately obese, adjusted for ethnicity), reduced mobility, active malignancy, major surgery within 6 weeks preceding first dose of study drug, post-partum within 12 weeks preceding first dose of study drug.
7. Women who are using estrogen-containing medication or hormone modulators (within 8 weeks pre-dose to 8 weeks post-dose of study drug).
8. Clinically significant cardiovascular disease.
9. Other conditions that substantially increase the risk of cardiovascular events by the discretion of the Investigator including, but not limited to: smoking, cocaine use, and uncontrolled hypertension.
10. Congenital or acquired bleeding disorders other than Glanzmann thrombasthenia.
11. Concurrent disease, treatment, medication, or abnormality in clinical laboratory tests that may pose additional risk.
12. Addiction or other diseases that prevent the participant from appropriately assessing the nature and scope of the clinical study or participating in study procedures.
13. Received any live vaccine within 4 weeks of enrollment or is planning to have a live vaccine during the study period.
14. Received investigational medication in another clinical study within 5 half-lives before administration of study drug.
15. Female participants who are pregnant or breastfeeding.

Part B Exclusion Criteria

1. Active severe infection or inflammation at the time of Screening or prior to the first dose of study drug.
2. History of clinically significant hypersensitivity associated with monoclonal antibody therapies.
3. Personal history of venous or arterial thrombosis or thromboembolic disease, with the exception of catheter-associated, superficial vein thrombosis.
4. Co-existing thrombophilic disorder, as determined by the presence of any of the below (or via historical results, where available):

   * Homozygous for Factor V Leiden gene mutation
   * Compound heterozygous for Factor V Leiden gene mutation
   * Prothrombin G20210A mutation
   * Antithrombin III, Protein C deficiency or Protein S deficiency with activity levels of ≤50% in participants with at least 1 second-degree relative with an unprovoked venous thromboembolism (VTE), or a first-degree relative with a minimally provoked VTE or at Investigator discretion for participants with an unknown family history
5. Family history of unprovoked venous thrombosis in first degree relative.
6. Has a positive test for HbsAg, HCV Ab, or HIV Ab at Screening with RNA level above the lower limit of detection. Participants with a positive test for HCV Ab may be included if they have a negative RNA test, consistent with cleared infection. Participants with an HIV RNA level lower than the limit of detection may be included.
7. Other conditions that substantially increase risk of thrombosis by the discretion of the investigator including, but not limited to: BMI >30 kg/m2 (moderately obese, adjusted for ethnicity), reduced mobility, active malignancy major surgery within 6 weeks preceding first dose of study drug, post-partum within 12 weeks preceding first dose of study drug.
8. Women who are using estrogen-containing medication or hormone modulators from 8 weeks prior to the first dose of study drug until 8 weeks after the last dose of study drug (see separate inclusion criterion for non-estrogen containing contraception requirement).
9. Clinically significant cardiovascular disease.
10. Other conditions that substantially increase risk of cardiovascular events by the discretion of the Investigator including, but not limited to: smoking tobacco products, cocaine use, uncontrolled hypertension and untreated hyperlipidemia.
11. Congenital or acquired bleeding disorders other than Glanzmann thrombasthenia.
12. Concurrent disease, treatment, medication, or abnormality in clinical laboratory tests that may pose additional risk.
13. Addiction or other diseases that prevent the participant from appropriately assessing the nature and scope of the clinical study or participating in study procedures.
14. Received any live vaccine within 4 weeks of enrollment or is planning to have a live vaccine during the study period.
15. Received investigational medication in another clinical study within 5 half-lives before administration of study drug.
16. Female participants who are pregnant (including a positive serum pregnancy test at Screening) or breastfeeding.

Ages: 18 Years to 67 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Estimated)
Dates: Start 2022-12-13 (Actual); Primary Completion 2027-08 (Estimated); Study Completion 2027-08 (Estimated)

PRIMARY OUTCOMES:
Part A: Safety as assessed by the incidence of treatment-emergent adverse events (TEAEs) | From baseline to Day 57
Part A: Safety as assessed by the changes in physical examinations, vital signs, clinical laboratory assessments, and ECG parameters | From baseline to Day 57
Part B: Safety as assessed by the incidence of treatment-emergent AEs | From baseline to Day 106/Early Termination (ET)/End of Study (EOS)
Part B: Safety as assessed by the changes in physical examinations, vital signs, clinical laboratory assessments, and ECG parameters | From baseline to Day 106/ET/EOS
Part B: Preliminary prophylactic effect of HMB-001 as assessed via Bleed frequency: annualized bleed rate (ABR) | From baseline to Day 106/ET/EOS
Part B: Preliminary prophylactic effect of HMB-001 as assessed via Bleed frequency: annualized treated bleed rate (ATBR) | From baseline to Day 106/ET/EOS
Part C: Safety as assessed by the incidence of treatment-emergent AEs | Day 99 to Day 687/Early Termination (ET)/ENdo of Study (EOS)
Part C: Safety as assessed by the changes in physical examinations, vital signs, clinical laboratory assessments, and ECG parameters | Day 99 to Day 687/Early Termination (ET)/ENdo of Study (EOS)
Part C: Preliminary prophylactic effect of HMB-001 as assessed via Bleed frequency: annual treated bleed rate (ATBR) and annualized bleed rate (ABR) | Day 99 to Day 687/Early Termination (ET)/ENdo of Study (EOS)

SECONDARY OUTCOMES:
Part A: Plasma concentrations of HMB-001 | From baseline to Day 57
Part A: Pharmacokinetics (PK) parameters: Maximum observed plasma concentration (Cmax) | From baseline to Day 57
Part A: PK parameters: Area under the curve from time zero to last quantifiable concentration (AUClast) | From baseline to Day 57
Part A: PK parameters: Area under the curve from time zero to extrapolated infinite time (AUCinf) | From baseline to Day 57
Part A: PK parameters: Time to reach maximum observed plasma concentration (Tmax) | From baseline to Day 57
Part A: Anti-drug antibody (ADA) formation | From baseline to Day 57
Part A: PD parameters: Maximum, mean increase in Coagulation factor VII (FVII) from baseline | From baseline to Day 57
Part A: PD parameters: Maximum, mean decrease from baseline in prothrombin time (PT) | From baseline to Day 57
Part A: PD parameters: Maximum, mean decrease from baseline in activated partial thromboplastin time (aPTT) | From baseline to Day 57
Part B: Plasma concentrations of HMB-001 | From baseline to Day 106/ET/EOS
Part B: PK parameters: Cmax | From baseline to Day 106/ET/EOS
Part B: PK parameters: AUClast | From baseline to Day 106/ET/EOS
Part B: PK parameters: AUCinf | From baseline to Day 106/ET/EOS
Part B: PK parameters: Tmax | From baseline to Day 106/ET/EOS
Part B: Preliminary prophylactic effect of HMB-001 as assessed by Subcategories of ABR, including, but not limited to spontaneous and impactful | From baseline to Day 106/ET/EOS
Part B: Preliminary prophylactic effect of HMB-001 as assessed by Bleed Severity (occurrence of severe bleeding events) | From baseline to Day 106/ET/EOS
Part B: Preliminary prophylactic effect of HMB-001 as assessed by the volume of transfusion product use | From baseline to Day 106/ET/EOS
Part B: Preliminary prophylactic effect of HMB-001 as assessed by the Volume of FVIIa use | From baseline to Day 106/ET/EOS
Part B: Preliminary prophylactic effect of HMB-001 as assessed by the Volume of red blood cell (RBC) transfusion | From baseline to Day 106/ET/EOS
Part B: Preliminary prophylactic effect of HMB-001 as assessed by the Iron Status: Mean change in hemoglobin from baseline | From baseline to Day 106/ET/EOS
Part B: Preliminary prophylactic effect of HMB-001 as assessed by the Iron Status: Mean change in ferritin and total iron from baseline | From baseline to Day 106/ET/EOS
Part B: ADA formation | From baseline to Day 106/ET/EOS
Part B: Changes from baseline in Euro Quality of life 5-Dimensions 5-Level (EQ-5D-5L) score | From Baseline to Day 85/End of Treatment (EOT)
Part B: Changes from baseline in Patient-Reported Outcomes Measurement Information System (PROMIS)-29 score | From Baseline to Day 85/End of Treatment (EOT)
Part B: Changes from baseline in Work Productivity and Activity Impairment (WPAI) score | From Baseline to Day 85/End of Treatment (EOT)
Part C: Plasma concentrations of HMB-001 | Day 99 to Day 687/Early Termination (ET)/ENdo of Study (EOS)
Part C: PK parameters: Cmax | Day 99 to Day 687/Early Termination (ET)/ENdo of Study (EOS)
Part C: PK parameters: AUClast | Day 99 to Day 687/Early Termination (ET)/ENdo of Study (EOS)
Part C: PK parameters: AUCinf | Day 99 to Day 687/Early Termination (ET)/ENdo of Study (EOS)
Part C: PK parameters: Tmax | Day 99 to Day 687/Early Termination (ET)/ENdo of Study (EOS)
Part C: Preliminary prophylactic effect of HMB-001 as assessed by Bleeding Events | Day 99 to Day 687/Early Termination (ET)/ENdo of Study (EOS)
Part C: Preliminary prophylactic effect of HMB-001 as assessed by Bleed Severity (occurrence of severe bleeding events) | Day 99 to Day 687/Early Termination (ET)/ENdo of Study (EOS)
Part C: Preliminary prophylactic effect of HMB-001 as assessed by the volume of transfusion product use | Day 99 to Day 687/Early Termination (ET)/ENdo of Study (EOS)
Part C: Preliminary prophylactic effect of HMB-001 as assessed by the Volume of FVIIa use | Day 99 to Day 687/Early Termination (ET)/ENdo of Study (EOS)
Part C: Preliminary prophylactic effect of HMB-001 as assessed by the Volume of red blood cell (RBC) transfusion | Day 99 to Day 687/Early Termination (ET)/ENdo of Study (EOS)
Part C: Preliminary prophylactic effect of HMB-001 as assessed by the Iron Status: Mean change in hemoglobin from baseline | Day 99 to Day 687/Early Termination (ET)/ENdo of Study (EOS)
Part C: Preliminary prophylactic effect of HMB-001 as assessed by the Iron Status: Mean change in ferritin and total iron from baseline | Day 99 to Day 687/Early Termination (ET)/ENdo of Study (EOS)
Part C: ADA formation | From baseline to Day 673/End of Treatment (EOT)
Part C: Changes from baseline in Euro Quality of life 5-Dimensions 5-Level (EQ-5D-5L) score | From baseline to Day 673/End of Treatment (EOT)
Part C: Changes from baseline in Patient-Reported Outcomes Measurement Information System (PROMIS)-29 score | From baseline to Day 673/End of Treatment (EOT)
Part C: Changes from baseline in Work Productivity and Activity Impairment (WPAI) score | From baseline to Day 673/End of Treatment (EOT)

CONTACTS AND LOCATIONS:
Locations (17):
- United States (5):
  - University of California, San Diego (UCSD) (Part B/C), La Jolla, California
  - Tulane University Medical Center (Part B/C), New Orleans, Louisiana
  - Mayo Clinic - Rochester (Part B/C), Rochester, Minnesota
  - Hemophilia Center of Western Pennsylvania (HCWP) (Part B/C), Pittsburgh, Pennsylvania
  - Washington Institute for Coagulation (Part B/C), Seattle, Washington
- University Hospital Leuven - Campus Gasthuisberg (Part B/C), Leuven, Belgium
- France (3):
  - AP-HP Hopital Bicetre (Part B/C), Le Kremlin-Bicêtre
  - AP-HM - Hopital de la Timone, Marseille
  - AP-HP Hopital Necker-Enfants Malades (Part B/C), Paris
- Italy (2):
  - Azienda Ospedaliero-Universitaria Careggi (Part B/C), Florence
  - Fondazione IRCCS Ca' Granda Ospedale Maggiore Policlinico di Milano (Part B/C), Milan
- Universitair Medisch Centrum Utrecht (Part B/C), Utrecht, Netherlands
- United Kingdom (5):
  - Queen Elizabeth Hospital Birmingham (Part B/C), Birmingham
  - Leeds Teaching Hospitals NHS Trust, Leeds
  - Richmond Pharmacology Ltd (Part A/B/C), London
  - Royal Free London NHS Foundation Trust (Part B/C), London
  - The Royal London Hospital (Part B/C), Whitechapel

IPD SHARING:
Plan to Share IPD: No